CLINICAL TRIAL: NCT06278545
Title: Randomized Phase II Trial Evaluating Modified FOLFIRINOX and Modified FOLFOX in the Treatment of Locally Advanced or Metastatic Small Bowel Adenocarcinoma
Brief Title: Trial Evaluating Modified FOLFIRINOX and Modified FOLFOX in the Treatment of Locally Advanced or Metastatic Small Bowel Adenocarcinoma
Acronym: FOLFORINOX SBA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MANFREDI PHRCK 2022
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced or Metastatic Small Bowel Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified FOLFIRINOX regimen D1=D15 (1 course every 14 days) (Experimental)
  Interventions: Drug: modified FOLFORINOX
- Modified FOLFOX regimen D1=D15 (1 course every 14 days) (Active Comparator)
  Interventions: Drug: Modified FOLFOX

INTERVENTIONS:
Drug: modified FOLFORINOX — One treatment every 14 days :
  * Irinotecan 180mg/m² as a 2-hour IV infusion
  * Oxaliplatin 85 mg/m² as a 2-hour IV infusion
  * Folinic acid 400 mg/m² as 2-hour IV infusion, in Y with oxaliplatin
  * 5-FU 2400 mg/m² as a continuous IV infusion over 46 hours
  Arms: Modified FOLFIRINOX regimen D1=D15 (1 course every 14 days)
Drug: Modified FOLFOX — One treatment every 14 days:
  * Oxaliplatin 85 mg/m by IV infusion over 2 hours
  * Folinic acid: 400 mg/m² or 200 mg/m² if laevorotatory form by IV infusion over 2 hours, in Y with oxaliplatin
  * 5FU bolus: 400 mg/m² per 10-minute IV infusion
  * 5 FU continuous 2400 mg/m² by IV infusion over 46 hours
  Arms: Modified FOLFOX regimen D1=D15 (1 course every 14 days)

SUMMARY:
Randomized, non-comparative, open-label, multi-centre Phase II study to evaluate modified FOLFIRINOX and modified FOLFOX in the locally advenced or metastatic small bowel adenocarcinoma.

The primary objective is to assess the percentage of patients alive without prograssion at 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the small intestine (duodenum, jejunum, ileum)
* Metastatic or locally advanced unresectable tumour with curative intent
* Patient who never received first-line chemotherapy
* Measurable lesion according to RECIST 1.1 criteria
* ECOG status < or = 2 for patients under 70 years, or 0 or 1 for patients over 70 years
* Life expectancy estimated at over 3 months
* Patient over 18 years of age
* Patient able to understand and sign the information and informed consent note
* Women of childbearing age and men who have sex with women of childbearing age must agree to use contraception during the trial treatment and for at least 9 months after stopping the experimental treatments.

Exclusion Criteria:

* MSI/dMMR tumor
* Adenocarcinoma of the ampulla of Vater
* Neutrophils < 1500/mm3, platelets < 100 000/mm3
* Hemoglobin < 9 g/dL, total bilirubin > 1.5x normal, alkaline phosphatase > 2.5x normal (or >5x normal if liver metastases), creatinine clearance > or = 40 ml/min. according to MDRD
* Hypokalaemia, hypomagnesaemia and hypocalcaemia below normal, and for calcaemia, it must be corrected before enrolment.
* Adjuvant chemotherapy completed less than 6 months ago
* History of myocardial infarction within the last 6 months, severe coronary artery disease or severe heart failure
* Severe renal failure
* Peripheral sensory neuropathy with functional discomfort
* Active and/or potentially severe infection or other uncontrolled conditions
* Treatment with a cytochrome P450 inhibitor within 4 weeks prior to the administration of the protocol treatment (refer to paragraph 8.3 "Contraindicated treatments" of the protocol)
* Patients currently undergoing treatment using St John's Wort
* Treatment with brivudine within 4 weeks prior to the administration of protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Assess the percentage of patients alive without progression | At 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France